CLINICAL TRIAL: NCT03412929
Title: A Clinical Evaluation of a Manuka-Honey Impregnated Dressing at Removing Necrotic Tissue From Chronic Foot and Ankle Wounds
Brief Title: A Clinical Evaluation of a Honey Impregnated Dressing at Removing Necrotic Tissue From Chronic Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R16-017
Record Dates: First submitted 2018-01-11; First posted 2018-01-29 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Wound Heal; Necrotic Tissue Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Honey Impregnated Dressing (Experimental): Honey Impregnated Dressing
  Interventions: Device: Honey Impregnated Dressing

INTERVENTIONS:
Device: Honey Impregnated Dressing — The investigational product being examined contains 100% Manuka honey and is ideal for difficult to dress wounds. The dressing provides a moist wound environment to help promote autolytic debridement. The dressing is ideal for partial or full thickness wounds with moderate-to-heavy drainage.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a honey-impregnated wound dressing at removing necrotic tissue in subjects with chronic foot or ankle wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Subject has a qualified chronic foot or ankle wound, sized 1cm2 to 25 cm2 for ≥ 4 weeks in duration
* Must have necrotic tissue at least 25% of wound area
* The wound type matches one of the indicated wounds listed on the product labeling:
* Leg ulcers
* Pressure ulcers
* Diabetic foot ulcers
* First and second degree burns
* Surgical wounds
* Trauma wounds
* Subject has adequate circulation as demonstrated by biphasic or triphasic Doppler waveform, consistent with adequate blood flow, within 3 months prior to study enrollment. If monophasic on exam, the non-invasive tests must display Ankle Brachial Index over 0.8 and no worse than mild disease on segmental pressures.
* Subject is likely to be compliant with instructions for case, such as following institutional standard of care directions, offloading, and keeping the wound area protected from environmental contaminants
* Type I/II diabetic subjects that meet the following criteria:
* Random blood glucose is less than 450 mg/dL within 30 days of the screening visit

Exclusion Criteria:

* Subject has a known sensitivity or allergy to honey based products, bee venom, or other ingredients in product
* The subject is breastfeeding, pregnant, or has intentions of becoming pregnant during the course of their study participation
* Wound duration ≥ 52 weeks
* The subject has a prognosis that indicated unlikely survival past the study period
* The subject is currently receiving dialysis
* Gangrene is present in the target wound
* Patient's wound is infected
* The subject's diagnosis indicates third degree burns
* The subject has received any treatment prior to study enrollment that may, in the opinion of an Investigator, affect the outcome of the study
* In the opinion of an Investigator, the subject is otherwise not suitable for study participation, such as the subject is likely to be non-compliant with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Illinois Foot & Ankle Specialists, Lake in the Hills, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Honey Impregnated Dressing
Started | 8
Completed | 5
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Necrotic Tissue
Description: The percent change in necrotic tissue will serve as the primary endpoint.
Time Frame: From initial date of application to weekly visits assessed up to 4 weeks.
Measure: Mean (95% Confidence Interval); unit: percent of necrotic tissue
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
percent of necrotic tissue | 40 [10 to 70]

2. Secondary Outcome: Wound Closure
Description: Percent of patients with 100% wound closure in each group
Time Frame: From initial date of application to weekly visits assessed up to 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Infections
Description: Number of infections in the wound sites will be recorded.
Time Frame: From initial date of application to weekly visits assessed up to 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Odor
Description: The odor score will be recorded using a scale of 1-4 with a score of 1 being pleasant odor to 4 being an unpleasant odor.
Time Frame: The odor score will be recorded at weekly visits over four weeks for each subject.
Population: Study staff reported scores of 0 when no odor was detectable.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
score on a scale
  Odor Score Initial Visit | 1 [1 to 3]
  Odor Score Final Visit | 1 [0 to 1]

5. Secondary Outcome: Pain Score
Description: The pain score will be recorded with a visual analog scale from 0-10. 0 is interpreted as no pain and 10 is the worst imaginable pain.
Time Frame: The pain score will be recorded at weekly visits over four weeks for each subject.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
score on a scale
  Pain Score Initial Visit | 0 [0 to 1]
  Pain Score Final Visit | 0 [0 to 0]

6. Secondary Outcome: Bates-Jensen Wound Assessment Tool Score
Description: The Bates-Jensen Wound Assessment tool score will be used to assess the wound's status. The Bates-Jensen Wound Assessment tool measures wound status. The wound size score ranges from 0 to 5. The wound depth score ranges from 0 to 5. The wound edge score ranges from 0 to 5. The wound undermining score ranges from 0 to 5. The necrotic tissue type score ranges from 1 to 5. The necrotic tissue amount ranges from 1 to 5. The exudate type score ranges from 1 to 5. The exudate amount score ranges from 1 to 5. The skin color surrounding wound score ranges from 1 to 5. The peripheral tissue edema score ranges from 1 to 5. The peripheral tissue induration score score ranges from 1 to 5. The granulation tissue score ranges from 1 to 5. The epithelialization score ranges from 1 to 5. The total score from these sub-scores added together is used as the total BWAT score. For all sub-score values, a value of 0 or 1 is a better outcome. The minimum total score is 9 and the maximum total score is 65.
Time Frame: The BWAT score will be recorded at weekly visits over fours weeks for each subject.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Honey Impregnated Dressing
Number analyzed (Participants) | 5
score on a scale
  BWAT Score Initial Visit | 35.4 [29.4 to 41.4]
  BWAT Score Final Visit | 23.6 [14.5 to 32.7]

ADVERSE EVENTS:
Time Frame: baseline to 4 weeks
Arm/Group | Honey Impregnated Dressing
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Honey Impregnated Dressing (N=8)
Swelling (Vascular disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03412929/Prot_SAP_000.pdf